CLINICAL TRIAL: NCT02206555
Title: Implementation of HIV Preexposure Prophylaxis With Antiretroviral Medications Among People at High Risk for HIV Infection: A Demonstration Project
Brief Title: PrEP Demonstration Project (PRELUDE Study)
Acronym: PRELUDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HEPP 1403; 14/098 (Other: St Vincent's Hospital HREC)
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: HIV
Keywords: HIV; prevention; prophylaxis; antiretroviral; biomedical; bio-behavioural; evaluation; demonstration study
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (TRUVADA) (Experimental): Homosexual men and heterosexual men and women at high risk of HIV infection
  Interventions: Drug: emtricitabine/tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: emtricitabine/tenofovir disoproxil fumarate
  Other Names: TRUVADA; FTC/TDF

SUMMARY:
Significant increases in HIV diagnoses among gay and other homosexually active men, in Australia and internationally, have been observed since the late 1990s. The levels of high HIV risk sexual practices among gay men have also increased, particularly unprotected anal intercourse (UAI). Nationally, over three quarters of the new HIV infections diagnosed annually are among men who have sex with men (MSM). The proportion of heterosexual men and women among those diagnosed with HIV annually has also increased in recent years. Despite successes in some situations, HIV transmission has not been adequately reduced by the prevention methods available to those at risk, such as education, condoms, and treatment of sexually transmitted infections (STIs).

The effectiveness of daily oral antiretroviral medications (ARVs) as preexposure prophylaxis of HIV (PrEP) has now been established by clinical trials in both heterosexual adults and homosexual men. Whether PrEP confers high rates of protection in real life situations and is a feasible strategy to implement still requires further investigation. Through its "HIV prevention strategy 2015: New era," NSW Health committed to consider how to most appropriately and efficiently implement PrEP in line with evidence. This commitment translated in the support to this PrEP demonstration project.

This demonstration project is designed to evaluate the off-label provision of daily combination of tenofovir disoproxil fumarate and emtricitabine (TDF/FTC, known as TRUVADA) as PrEP to a sample of sero-negative individuals at high risk for HIV infection in clinical settings in New South Wales. The project will inform policy development regarding primary HIV prevention with PrEP.

This is an open-label, single-arm treatment evaluation study. All consenting and eligible HIV negative participants will receive TRUVADA prescribed for daily administration orally. At each followup visit, the following procedures will be conducted: clinical evaluations/ procedures, laboratory evaluations/ procedures, testing for HIV, STIs, hepatic and renal function, assessment for adherence to the prescribed medication, side effects, eligibility for next TRUVADA prescription, and willingness to continue on PrEP.

As a study requirement, participants will be offered a self-administered assessment of behaviour, lifestyle and attitudes which will be conducted ideally within two and no more than seven days of the clinic visit in the participant's private space.

Analyses will include: the feasibility of PrEP delivery, adherence to the study medication, safety and tolerability, the effects of PrEP use on behavior, and statistical analyses of the risk of HIV seroconversion.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative at enrollment (per algorithm provided in protocol)
* At high and ongoing risk for acquiring HIV infection (per algorithm provided in protocol)
* Aged 18 years or over
* Resident of NSW (or elsewhere in Australia if they visit NSW with sufficient frequency to allow participation)
* Medicare eligible (to have Medicare coverage for the standard-of-care services)
* Willing and able to provide informed consent
* Willing and able to take part in all required study procedures
* Proficiency in written and spoken English (necessary to complete attitude, behavioural and lifestyle surveys)

Exclusion Criteria:

* HIV-1 infected or has symptoms consistent with acute viral infection (If HIV positive status is not confirmed by testing, delay starting PrEP for at least one month and reconfirm negative HIV-1 status).
* Having an estimated creatinine clearance (glomerular filtration rate [GFR]) <60ml/min
* Having or developing clinical symptoms suggestive of lactic acidosis or pronounced hepatotoxicity (including nausea, vomiting, unusual or unexpected stomach discomfort, and weakness)
* Concurrently taking a nephrotoxic agent (e.g., high-dose non-steroidal anti-inflammatory drugs / NSAIDs)
* Allergic to tenofovir disoproxil fumarate and/or emtricitabine (based on self-report or recorded)
* Concurrently taking prescribed products containing emtricitabine or tenofovir disoproxil fumarate including ATRIPLA®, COMPLERA®, EMTRIVA, STRIBILD®, VIREAD; other drugs containing lamivudine; HEPSERA
* Mental health issues, memory loss or other cognitive impairment or intellectual disability that may compromise participant safety and/or regimen adherence
* Factors or conditions that may compromise a participant's retention in the study (incarceration, planned relocation or potential absence from NSW for a period of 3 months or longer during the course of the study)
* Unwilling to adhere to any of the required study procedures
* Currently breastfeeding

Note: Safety for infants exposed to TRUVADA during pregnancy is not fully assessed but no harm has been reported. Therefore, planning to become pregnant or currently being pregnant is not an exclusion criterion for this study. However, women who are pregnant should learn about the risks and benefits of TRUVADA to reduce the risk of acquiring HIV during their pregnancy. Site investigators will review the risks and benefits of TRUVADA and of potential HIV infection with pregnant women and women who plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Time to accrual | Approximately 18 months
  Time to accrual of 300 person-years of follow-up on TRUVADA. Each participant will receive TRUVADA for a maximum of 12 months, and will be followed for an additional three months after discontinuation. (Primary endpoint: feasibility of the process of PrEP delivery in health care settings in NSW)
Seroconversion-free time on PrEP | Approximately 18 months
  Seroconversion-free time on PrEP (Primary endpoint: feasibility of the process of PrEP delivery in health care settings in NSW)
Time to TRUVADA discontinuation | Approximately 18 months
  Time to TRUVADA discontinuation (primary endpoint: adherence)
Prescribed doses taken | Approximately 18 months
  Percentage of prescribed doses taken orally in the prescribed period (primary endpoint: adherence)
Incidents of HIV seroconversion | Approximately 24 months
  Incidence of HIV seroconversion among study participants during the course of their study participation and in six months following PrEP discontinuation (primary endpoint: safety and side effects)
Incidents of rectal gonorrhea and chlamydia | Approximately 18 months
  New rectal gonorrhoea and chlamydia infections (primary endpoint: behavioral effects of PrEP use)
Serious adverse reactions | Approximately 18 months
  (primary endpoint: safety and side effects)
Adverse events | Approximately 18 months
  Any adverse events leading to interruption or discontinuation of the study product (TRUVADA) (primary endpoint: safety and side effects)

CONTACTS AND LOCATIONS:
Overall Officials: Iryna Zablotska, MD, MPH, PhD, Study Chair — Kirby Institute
Locations (5):
- Australia (5):
  - RPA Sexual Health, Camperdown, New South Wales
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St Vincent's Hospital HIV, Immunology and Infectious Disease Unit, Darlinghurst, New South Wales
  - Western Sydney Sexual Health Centre, Parramatta, New South Wales
  - Sydney Sexual Health Centre, Sydney, New South Wales

REFERENCES:
- [Derived] Vaccher SJ, Marzinke MA, Templeton DJ, Haire BG, Ryder N, McNulty A, Foster R, Grulich AE, Zablotska IB; PRELUDE Study Team; NSW HIV Prevention Partnership Project. Predictors of Daily Adherence to HIV Pre-exposure Prophylaxis in Gay/Bisexual Men in the PRELUDE Demonstration Project. AIDS Behav. 2019 May;23(5):1287-1296. doi: 10.1007/s10461-018-2353-5. PMID 30523489
- [Derived] Vaccher SJ, Gianacas C, Templeton DJ, Poynten IM, Haire BG, Ooi C, Foster R, McNulty A, Grulich AE, Zablotska IB; PRELUDE Study Team. Baseline Preferences for Daily, Event-Driven, or Periodic HIV Pre-Exposure Prophylaxis among Gay and Bisexual Men in the PRELUDE Demonstration Project. Front Public Health. 2017 Dec 15;5:341. doi: 10.3389/fpubh.2017.00341. eCollection 2017. PMID 29326917
- [Derived] Vaccher S, Grulich A, McAllister J, Templeton DJ, Bloch M, McNulty A, Holden J, Poynten IM, Prestage G, Zablotska I; PRELUDE Study Team. Protocol for an open-label, single-arm trial of HIV pre-exposure prophylaxis (PrEP) among people at high risk of HIV infection: the NSW Demonstration Project PRELUDE. BMJ Open. 2016 Jun 20;6(6):e012179. doi: 10.1136/bmjopen-2016-012179. PMID 27324719